CLINICAL TRIAL: NCT00270647
Title: Physicians' Health Study II: Trial of Vitamins in the Chemoprevention of Cancer, CVD, and Eye Disease
Brief Title: Physicians' Health Study II
Acronym: PHS II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, John Michael Gaziano, MD, Physician, Brigham and Women's Hospital; Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: CDR0000448630; BWH-1999-P-003315; BWH-1999-P-003318; BWH-83-00405; R01CA097193 (NIH)
Record Dates: First submitted 2005-12-27; First posted 2005-12-28 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Cancer; Prostate Cancer; Colorectal Cancer; Cardiovascular Disease; Eye Disease; Cognitive Decline
Keywords: cancer; prostate cancer; colorectal cancer; cardiovascular disease; eye disease; cognitive decline
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Cardiovascular Diseases; Eye Diseases; Cognitive Dysfunction | interventions — Vitamin E; Ascorbic Acid; Geritol; beta Carotene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin E (Experimental): Active or placebo vitamin E
  Interventions: Dietary Supplement: Vitamin E
- Vitamin C (Experimental): Active or placebo vitamin C
  Interventions: Dietary Supplement: Vitamin C
- Multivitamin (Experimental): Active or placebo multivitamin
  Interventions: Dietary Supplement: Multivitamin
- Beta-carotene (Experimental): Active or placebo beta-carotene
  Interventions: Dietary Supplement: Beta-carotene

INTERVENTIONS:
Dietary Supplement: Vitamin E — 400 IU synthetic alpha-tocopherol or its placebo on alternate days (provided by BASF)
  Arms: Vitamin E
Dietary Supplement: Vitamin C — 500 mg synthetic ascorbic acid or its placebo daily (provided by BASF)
  Arms: Vitamin C
Dietary Supplement: Multivitamin — Centrum Silver or its placebo daily (provided by Pfizer (formerly Wyeth, American Home Products, and Lederle))
  Arms: Multivitamin
Dietary Supplement: Beta-carotene — 50 mg Lurotin or placebo on alternate days (provided by BASF)
  Arms: Beta-carotene

SUMMARY:
The use of vitamin E, vitamin C, beta carotene, and/or multivitamins may keep cancer, cardiovascular disease, eye diseases, or cognitive decline from occurring. This randomized clinical trial studied vitamin E, vitamin C, beta carotene, and/or multivitamins to see how well they work compared with placebos in preventing cancer, cardiovascular disease, eye disease, and cognitive decline in male doctors aged 50 years and older.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether vitamin E every other day reduces the risk of developing prostate cancer in older healthy male physicians.
* To determine whether daily vitamin C and/or a multivitamin reduces the risk of total cancer in these participants.
* To determine whether vitamin E every other day, vitamin C daily, or a multivitamin daily reduces the risk of major cardiovascular events in these participants.

Secondary

* To determine whether vitamin E and/or multivitamins reduce the risk of developing total cancer, colon cancer, and colon polyps in these participants.
* To determine whether vitamin E, vitamin C, or multivitamins reduce the risk of myocardial infarction and stroke in these participants.
* To determine whether vitamin E, vitamin C, or multivitamins reduce the risk of age-related macular degeneration or cataract in these participants.
* To determine whether vitamin E, vitamin C, or multivitamins reduce the risk of early cognitive decline in participants aged 65 and over.

The Physicians' Health Study II was a randomized, double-blind, placebo-controlled, factorial trial that began in 1997 and ended in 2011. It was designed to test four supplements -- (1) alternate-day vitamin E (400 international units of synthetic alpha-tocopherol) or its placebo; (2) daily vitamin C (500 mg synthetic ascorbic acid) or its placebo; (3) a daily multivitamin (Centrum Silver) or its placebo; and (4) alternate-day beta carotene (50 mg Lurotin) or its placebo -- in the prevention of cancer, cardiovascular disease, eye disease, and early cognitive decline among 14,641 male physicians aged 50 years or older. Participants were randomly assigned in a 2x2x2x2 factorial trial to receive combinations of the four active supplements or their placebos. Pills and/or packaging were provided by BASF Corporation, Pfizer (formerly Wyeth, American Home Products, and Lederle), and DSM Nutritional Products (formerly Roche Vitamins).

The beta-carotene component was discontinued on March 8, 2003; the vitamin E and vitamin C components ended as scheduled on August 31, 2007; and the multivitamin component ended on June 1, 2011.

ELIGIBILITY:
INCLUSION CRITERIA

1. DISEASE CHARACTERISTICS:

   * Healthy male physicians practicing in the United States
   * Prior participation in the Physicians' Health Study I allowed
2. PATIENT CHARACTERISTICS:

   * Aged 50 years and over
   * No history of serious illness that would preclude study participation
   * No history of significant adverse events (e.g., rash or allergic reaction) attributed to study agents
3. PRIOR CONCURRENT THERAPY:

   * No other concurrent vitamin and/or multivitamin supplementation
   * No concurrent vitamin K-depleting anticoagulants (e.g., warfarin)

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14641 (Actual)
Dates: Start 1997-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Prostate cancer | Ongoing
Total cancer | Ongoing
Major cardiovascular events | Ongoing

SECONDARY OUTCOMES:
Cataract | Ongoing
Age-related macular degeneration | Ongoing
Early cognitive decline | Ongoing
Myocardial infarction | Ongoing
Stroke | Ongoing
Colorectal cancer | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: J. Michael Gaziano, MD, MPH, Principal Investigator — Brigham and Women's Hospital

REFERENCES:
- [Background] Christen WG, Gaziano JM, Hennekens CH. Design of Physicians' Health Study II--a randomized trial of beta-carotene, vitamins E and C, and multivitamins, in prevention of cancer, cardiovascular disease, and eye disease, and review of results of completed trials. Ann Epidemiol. 2000 Feb;10(2):125-34. doi: 10.1016/s1047-2797(99)00042-3. PMID 10691066
- [Result] Gaziano JM, Glynn RJ, Christen WG, Kurth T, Belanger C, MacFadyen J, Bubes V, Manson JE, Sesso HD, Buring JE. Vitamins E and C in the prevention of prostate and total cancer in men: the Physicians' Health Study II randomized controlled trial. JAMA. 2009 Jan 7;301(1):52-62. doi: 10.1001/jama.2008.862. Epub 2008 Dec 9. PMID 19066368
- [Result] Sesso HD, Buring JE, Christen WG, Kurth T, Belanger C, MacFadyen J, Bubes V, Manson JE, Glynn RJ, Gaziano JM. Vitamins E and C in the prevention of cardiovascular disease in men: the Physicians' Health Study II randomized controlled trial. JAMA. 2008 Nov 12;300(18):2123-33. doi: 10.1001/jama.2008.600. Epub 2008 Nov 9. PMID 18997197
- [Result] Christen WG, Glynn RJ, Sesso HD, Kurth T, Macfadyen J, Bubes V, Buring JE, Manson JE, Gaziano JM. Vitamins E and C and medical record-confirmed age-related macular degeneration in a randomized trial of male physicians. Ophthalmology. 2012 Aug;119(8):1642-9. doi: 10.1016/j.ophtha.2012.01.053. Epub 2012 Apr 13. PMID 22503302
- [Result] Christen WG, Glynn RJ, Sesso HD, Kurth T, MacFadyen J, Bubes V, Buring JE, Manson JE, Gaziano JM. Age-related cataract in a randomized trial of vitamins E and C in men. Arch Ophthalmol. 2010 Nov;128(11):1397-405. doi: 10.1001/archophthalmol.2010.266. PMID 21060040
- [Result] Grodstein F, Kang JH, Glynn RJ, Cook NR, Gaziano JM. A randomized trial of beta carotene supplementation and cognitive function in men: the Physicians' Health Study II. Arch Intern Med. 2007 Nov 12;167(20):2184-90. doi: 10.1001/archinte.167.20.2184. PMID 17998490
- [Derived] Juraschek SP, Gaziano JM, Glynn RJ, Gomelskaya N, Bubes VY, Buring JE, Shmerling RH, Sesso HD. Effects of vitamin C supplementation on gout risk: results from the Physicians' Health Study II trial. Am J Clin Nutr. 2022 Sep 2;116(3):812-819. doi: 10.1093/ajcn/nqac140. PMID 35575611
- [Derived] Rautiainen S, Gaziano JM, Christen WG, Bubes V, Kotler G, Glynn RJ, Manson JE, Buring JE, Sesso HD. Effect of Baseline Nutritional Status on Long-term Multivitamin Use and Cardiovascular Disease Risk: A Secondary Analysis of the Physicians' Health Study II Randomized Clinical Trial. JAMA Cardiol. 2017 Jun 1;2(6):617-625. doi: 10.1001/jamacardio.2017.0176. PMID 28384735
- [Derived] Wang L, Sesso HD, Glynn RJ, Christen WG, Bubes V, Manson JE, Buring JE, Gaziano JM. Vitamin E and C supplementation and risk of cancer in men: posttrial follow-up in the Physicians' Health Study II randomized trial. Am J Clin Nutr. 2014 Sep;100(3):915-23. doi: 10.3945/ajcn.114.085480. Epub 2014 Jul 9. PMID 25008853
- [Derived] Grodstein F, O'Brien J, Kang JH, Dushkes R, Cook NR, Okereke O, Manson JE, Glynn RJ, Buring JE, Gaziano M, Sesso HD. Long-term multivitamin supplementation and cognitive function in men: a randomized trial. Ann Intern Med. 2013 Dec 17;159(12):806-14. doi: 10.7326/0003-4819-159-12-201312170-00006. PMID 24490265
- [Derived] Christen WG, Glynn RJ, Manson JE, MacFadyen J, Bubes V, Schvartz M, Buring JE, Sesso HD, Gaziano JM. Effects of multivitamin supplement on cataract and age-related macular degeneration in a randomized trial of male physicians. Ophthalmology. 2014 Feb;121(2):525-34. doi: 10.1016/j.ophtha.2013.09.038. Epub 2013 Nov 20. PMID 24268861
- [Derived] Gaziano JM, Sesso HD, Christen WG, Bubes V, Smith JP, MacFadyen J, Schvartz M, Manson JE, Glynn RJ, Buring JE. Multivitamins in the prevention of cancer in men: the Physicians' Health Study II randomized controlled trial. JAMA. 2012 Nov 14;308(18):1871-80. doi: 10.1001/jama.2012.14641. PMID 23162860
- [Derived] Sesso HD, Christen WG, Bubes V, Smith JP, MacFadyen J, Schvartz M, Manson JE, Glynn RJ, Buring JE, Gaziano JM. Multivitamins in the prevention of cardiovascular disease in men: the Physicians' Health Study II randomized controlled trial. JAMA. 2012 Nov 7;308(17):1751-60. doi: 10.1001/jama.2012.14805. PMID 23117775